CLINICAL TRIAL: NCT05037877
Title: An Exploratory Investigation of Dietary Supplementation and Its Effect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HUM Nutrition, Inc. (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20220HUM
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Quality of Life

STUDY DESIGN:
Intervention Model Description: This will be a 2-arm randomized, double-blinded, placebo-controlled study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): HUM supplement - 1 capsule per day
  Interventions: Dietary Supplement: HUM supplement
- Placebo group (Placebo Comparator): Placebo supplement - 1 capsule per day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: HUM supplement — HUM supplement - 1 capsule per day
  Arms: Intervention group
Dietary Supplement: Placebo — Placebo supplement - 1 capsule per day
  Arms: Placebo group

SUMMARY:
The primary objective of this study is to understand if the test product (HUM supplement) improve symptoms experienced.

DETAILED DESCRIPTION:
This will be a 2-arm randomized, double-blinded, placebo-controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Willing to maintain the current dietary pattern, activity level, and stable body weight for the duration of the study
* Must be in good health (don't report any medical conditions asked in the screening questionnaire)
* Willing and able to provide written informed consent

Exclusion Criteria:

* Allergies to any test product ingredients
* Any other severe chronic disease
* Pregnant, want to become pregnant for the duration of the study, or who are breastfeeding
* Participating in an investigational health product research study

Ages: 38 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Quality of life improvements [Time Frame: Baseline to 8 weeks) | 8 week
  Survey-based assessment (0-5 scale) with higher scores representing an improved outcome

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Mitschke, Principal Investigator — Citruslabs
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No